CLINICAL TRIAL: NCT05329129
Title: PROSPECTIVE OBSERVATIONAL SPINE FUSION REGISTRY FOR OssDsign® BONE GRAFT SUBSTITUTES IN REAL WORLD CLINICAL PRACTICE
Brief Title: OssDsign® Spine Registry Study ("Propel")
Status: Recruiting | Type: Observational
Sponsor: OssDsign (Industry)
Responsible Party: Sponsor
Other Study IDs: OSD202101
Record Dates: First submitted 2022-03-22; First posted 2022-04-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis
Keywords: Synthetic bone grafts; Degenerative Disc Disease; Bone fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: OssDsign® Catalyst — An osteoconductive, resorbable, porous, 100 % nano synthetic calcium phosphate bone void filler

SUMMARY:
The purpose of this multi-center, prospective, observational registry is to gather information on the clinical outcomes and real-world use of commercially available bone graft substitutes manufactured by OssDsign® AB, in patients who require spine fusion.

DETAILED DESCRIPTION:
This multi-center study (up to 15 US study sites) is a post market, prospective, observational spine fusion registry. The outcomes of patients undergoing spine fusion with OssDsign® bone grafts will be documented and evaluated for the purposes of post market clinical follow up as part of OssDsign® post market surveillance activities. The length of study duration and number to be recruited is open-ended but initially a target of 450 subjects will be recruited and followed up for a period of 24 months ± 90 days after their index surgery in which an OssDsign® bone graft has been implanted.

ELIGIBILITY:
* The patient has been diagnosed as a candidate for spinal fusion surgery for which the surgeon has decided an OssDsign® bone graft is appropriate.
* The patient is ≥21 years old.
* The patient is, in the investigator's opinion, psychosocially, mentally, and physically able to fully comply with this protocol, including the post-operative regimen, required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent
* The patient is willing and able to participate in post- operative clinical and radiographic follow up evaluations for 2 years.

Exclusion Criteria:

* Patients not meeting all of the inclusion criteria

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with as a candidate for spinal fusion surgery
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2027-03-23 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of bone fusion | 12 months ± 60 days post-operative examination
  Assessment of the rate of bone fusion via Computerized Tomography (CT)/x-ray based on evidence of continuous bone bridging from the superior to the inferior vertebral body at the target level.

SECONDARY OUTCOMES:
Quality of Life Questionnaire: Oswestry Disability Index | Up to 4 months, 6, 12 and 24 months
  A questionnaire used to measure a patient's permanent functional disability scored 0-4, (no disability) to 35-50, (completely disabled).
Quality of Life Questionnaire: Neck Disability Index (NDI) | Up to 4 months, 6, 12 and 24 months
  A self-reported questionnaire to determine how pain affects everyday life and assess the level of disability and scored from 0 (no disability) to 50 (complete disability).
Quality of Life Questionnaire: Visual Analog Scale (VAS) | Up to 4 months, 6, 12 and 24 months
  A self rated pain scale from 0 (no pain) to 10 (worst imaginable pain)
Quality of Life Questionnaire: Short Form 36 (SF-36) | Up to 4 months, 6, 12 and 24 months
  A Questionnaire used to measure the impact of clinical and social interventions using eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability
Neurological Function | Up to 4 months, 6, 12 and 24 months
  All subjects will be assessed for sensory, reflex, and muscle strength (motor) by the clinician
Presence of bone fusion | 6, 12 and 24 months
  All subjects will undergo x-ray evaluation to include AP and neutral lateral views pre-operatively. At post-operative visits AP and neutral lateral x-rays, plus flexion and extension x-rays (if standard care) taken with the subject standing up and/or a CT scan taken.
Safety review of device related AE's | Throughout study, 24 months
  Review of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Marshall, Study Director — OssDsign
Locations (13):
- United States (13):
  - Community Health Partners Neuroscience, Fresno, California
  - San Diego Neurosurgery, San Diego, California
  - Orthopedic Associates of Hartford, Hartford, Connecticut
  - Central Connecticut Neurosurgery and Spine, New Britian, Connecticut
  - Yale Center for Clinical Investigation, Yale School of Medicine, New Haven, Connecticut
  - Minimally Invasive Spine Center of South Florida, Miami, Florida
  - Foundation for Orthopaedic Research and Education, Tampa, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Carle Foundation Hospital, NeuroScience Institute, Urbana, Illinois
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - OrthoBethesda Research Foundation, Bethesda, Maryland
  - Twin Cities Orthopedics, Edina, Minnesota
  - University Orthopedics Center, State College, Pennsylvania